CLINICAL TRIAL: NCT04617041
Title: Assessment of DAFILON® Suture Material for Skin Closure: A Prospective, Multicentric, International, Single-arm, Observational Study in Daily Practice
Brief Title: Assessment of DAFILON® Suture Material for Skin Closure
Acronym: SKINDA
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1909
Record Dates: First submitted 2020-10-20; First posted 2020-11-05 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Laceration of Skin; Injury Skin
Keywords: Non-absorbable suture; Skin closure; Surgical site infection; Wound dehiscence
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
In this non-interventional study (NIS) a polyamide non-absorbable suture (Dafilon®) will be evaluated for skin closure in adult and pediatric patients. The aim of the study is to collect clinical data on the performance of Dafilon® for skin closure. The results of this study will generate further clinical evidence for the use and the benefit of a non-absorbable surgical suture material produced from polyamide. Furthermore, the proactive collection of clinical data for Dafilon® suture will support the maintenance of the suture material on the market, so that in the future other patients can receive the suture material for skin closure.

ELIGIBILITY:
Inclusion:

* Written informed consent is available
* Patients undergoing skin closure with Dafilon®
* Small linear minimally contaminated incision/laceration in the trunk or extremities

Exclusion:

* Emergency surgery
* Pregnancy
* Facial lacerations or incisions
* Visible dirt in the wounds
* Nonlinear shape
* Patient taking medication that might affect wound healing
* Patient with hypersensitivity or allergy to the suture material

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: adult patients and children
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Combination of Surgical Site Infection (SSI) and Wound Dehiscence | until suture removal 10±5 days postoperatively.
  The hypotheses of the current study is that the combined endpoint which consists of the sum of the wound dehiscence and SSI rate will not be inferior to the rate of 13% published by Sajid M. S. et al., 2014 [Systematic review of absorbable vs non-absorbable sutures used for the closure of surgical incisions. World J Gastrointest Surg 2014 27;6(12): 241-247]

SECONDARY OUTCOMES:
Individual rate of surgical site infection (SSI) at discharge | until day of discharge (approximately 1-2 days postoperatively)
  Incidence of postoperative surgical site infections, SSI (A1: Superficial incisional site infections and A2: Deep incisional surgical site infections) (efficacy parameter) Surgical Site Infection (SSI) is defined according to the definition of the US Centres for Disease Control and Prevention (CDC).
Individual rate of surgical site infection (SSI) at postoperative Examination | 10±5 days postoperatively
  Incidence of postoperative surgical site infections, SSI (A1: Superficial incisional site infections and A2: Deep incisional surgical site infections) (efficacy parameter) Surgical Site Infection (SSI) is defined according to the definition of the US Centres for Disease Control and Prevention (CDC).
Individual dehiscence rate at discharge | until day of discharge (approximately 1-2 days postoperatively)
  Incidence of wound dehiscence (skin) in postoperative course
Individual dehiscence rate at postoperative Examination | 10±5 days postoperatively
  Incidence of wound dehiscence (skin) in postoperative course
Adverse events | until 10±5 days postoperatively
  Rates of postoperative complications such as tissue reaction or inflammation, seroma, abscess formation, hematoma, granuloma, bleeding, suture removal or re-suturing in postoperative course
Progress of Wound healing | until day of discharge (approximately 1-2 days postoperatively), 10±5 days post operatively and at follow-up visit
  This parameter will be noted using the Visual Analogue Scale (VAS) which states "0" at one end representing "worst wound healing" and "10" at the opposite end representing "excellent wound healing". The values are compared over postoperative period.
Progress of Cosmetic result | at 10±5 days (suture removal) and at optional follow-up visit
  Overall patient and observer satisfaction with the scar using the Patient and Observer Scar Assessment Scale (POSAS). Cosmetic result and the scar will be evaluated by the patient and the physician. Patient will rate the cosmetic outcome in six categories (Pain, Itching, Color of scar, Stiffness of scar, thickness and irregularity of scar) on a 1 to 10 points scale each. The physician will use the Observer component, rating vascularization, pigmentation, thickness, relief and pliability of the scar on a 1 to 10 points scale each. The categories are added to a total POSAS score of 11 (minimum) to 110 points (maximum). The values are compared over postoperative period.
Rate of hypertrophic scar | 10±5 days postoperatively (suture removal)
  A hypertrophic scar is a cutaneous condition characterized by deposits of excessive amounts of collagen which gives rise to a raised scar, but not to the degree observed with keloids. [wikipedia]
Rate of keloid scar | 10±5 days postoperatively (suture removal)
  Keloidal scar is the formation of a type of scar which, depending on its maturity, is composed mainly of either type III (early) or type I (late) collagen. It is a result of an overgrowth of granulation tissue (collagen type 3) at the site of a healed skin injury which is then slowly replaced by collagen type 1. Keloids should not be confused with hypertrophic scars, which are raised scars that do not grow beyond the boundaries of the original wound. [wikipedia]
Progress of Pain: Visual Analogue Scale (VAS) | until day of discharge (approximately 1-2 days postoperatively) and 10±5 days postoperatively
  This parameter will be noted using the Visual Analogue Scale (VAS) which state "0" at one end representing "no pain" and "100" at the opposite end representing "heavy pain". The values are compared over postoperative period.
Progress of Satisfaction: Visual Analogue Scale (VAS) | until day of discharge (approximately 1-2 days postoperatively) and 10±5 days postoperatively
  This parameter will be noted using the Visual Analogue Scale (VAS) which state "0" at one end representing "very poor" and "100" at the opposite end representing "excellent". The values are compared over postoperative period.
Assessment of the handling of the suture material | intra-operatively
  Assessment of the handling of the suture material intra-operatively using a questionnaire including different dimensions (knot security, tensile strength, knot run down, tissue drag, stiffness, etc.) with 5 evaluation levels (excellent, very good, good, satisfied, poor)
Length of hospital stay | until day of discharge (approximately 1-2 days postoperatively)
  Number of days between date of surgery and date of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Guillermo López Paredes, Dr., Principal Investigator — Hospital Vall D'Hebrón, Barcelona
Locations (2):
- Klinikum Landkreis Tuttlingen, Dept. General Surgery, Tuttlingen, Baden-Wurttemberg, Germany
- Hospital Universitario Vall d'Hebron, Barcelona, Spain